CLINICAL TRIAL: NCT04749654
Title: EFFECTS OF SPACE MAINTAINERS ON THE SALIVARY pH, FLOW RATE, STREPTOCOCCUS MUTANS AND LACTOBACILLUS CARRIAGE: AN IN VİVO STUDY
Brief Title: SPACE MAINTAINERS EFFECTS ON ORAL MİCROFLORA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, esra kizilci, DDS. PhD. Assistant Prof. Dr, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 149-3
Record Dates: First submitted 2020-11-16; First posted 2021-02-11 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-01

CONDITIONS: Orthodontic Appliance Complication; Lactobacillus Infection; Dental Caries in Children; Streptococcus, Other Specified Group
Keywords: Space maintainers; Streptococcus mutans; Lactobacillus; Salivary flow; Salivary pH

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fixed space maintainers (Experimental): band-and-loop type fixed space maintainers were applied
  Interventions: Other: The Salivary pH measured; Other: The saliva flow rate was measured; Other: Streptococcus mutans and Lactobacillus counts in saliva were measured
- Removable space maintainers (Experimental): All removable space maintainers were produced of an acrylic base and retention elements that were a vestibule arch, (Adam's and C clasps).
  Interventions: Other: The Salivary pH measured; Other: The saliva flow rate was measured; Other: Streptococcus mutans and Lactobacillus counts in saliva were measured

INTERVENTIONS:
Other: The Salivary pH measured — The saliva samples were obtained at 10-12 a.m. from all children. The saliva was collected into plastic cylinders and the salivary pH was measured with a pH meter (Compact pH meter B-212 twin pH, HORIBA, Osaka, Japan).
Other: The saliva flow rate was measured — The saliva flow rate was estimated by during the first 30 s of paraffin chewing. The saliva was collected into plastic cylinders for a period of 5 minutes. Afterward, the saliva were weighed with a in a precision balance (Mettler PC 400, Zurich, Switzerland) and the flow rate was computed in gms/ml.
Other: Streptococcus mutans and Lactobacillus counts in saliva were measured — The saliva samples were obtained according to described above. Numbers of colony-forming units (CFU) of S. mutans were counted on TSY20B agar and Lactobacilli were counted on Rogosa agar.

SUMMARY:
Space maintainers are used to preserve the space after premature loss of teeth but they could effect some factors that play a role in caries formation. The research aimed to assess the impacts of removable and fixed space maintainers on the salivary pH, flow rate, and Streptococcus mutans, Lactobacillus carriage.

DETAILED DESCRIPTION:
Although the usage of space maintainers can reduce the severity of problems that arise from the early loss of teeth, there are concerns regarding the impact of fixed and removable appliances on factors that can lead to dental caries. All space maintainer appliances are plaque retentive since bands and brackets increase the retention of plaque and food on tooth surfaces, reduce the clearance of plaque by saliva and make conventional oral hygiene for plaque removal more difficult, therefore, they may cause caries development.Space maintainers can favor caries formation by changing the oral microflora. patients aged between 4-10 years, each of whom had an indication for a fixed (n=19) or removable space maintainer (n=19), were enrolled in this research. The salivary pH, saliva flow rate, Streptococcus mutans and Lactobacillus counts in saliva were measured just prior to the application of space maintainers (baseline-T0) and in the course of the follow-up; at the 1st (T1), 3rd (T2), and 6th (T3) months. The Wilcoxon, Mann-Whithney U test and Friedman tests were used for statistical analyses.

ELIGIBILITY:
Inclusion Criteria:

* The present research was conducted on 38 patients aged between 4-10 years, each of whom had an indication for a fixed or removable space maintainer.

Exclusion Criteria:

* Patients with a medical history that could influence microorganism carriage, including systemic disease, immunosuppression and the usage of antibiotics in the preceding 15 days, were excluded from the research

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 38 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2013-07 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
FOR FıXED SPACE MAıNTAıNERS: CHANGES ON THE SALIVARY pH WERE MEASURED | baseline-1st month measure assessing change
  Salivary pH was measured by pH meter (pH= -log hydrogen ion)
FOR FıXED SPACE MAıNTAıNERS: CHANGES ON THE SALIVARY STREPTOCOCCUS MUTANS COUNTS WERE MEASURED | baseline-1st month measure assessing change
  Strep. mutans were counted by numbers of colony-forming units (CFU) per ml (milliliter)
FOR FıXED SPACE MAıNTAıNERS: CHANGES ON THE SALIVARY FLOW RATE WERE MEASURED | baseline-1st month measure assessing change
  Saliva flow rate was computed in ml/ min
FOR FıXED SPACE MAıNTAıNERS: CHANGES ON THE LACTOBACILLUS COUNTS WERE MEASURED | baseline-1st month measure assessing change
  Lactobacilli were counted by numbers of colony-forming units (CFU) per ml (milliliter)
FOR FıXED SPACE MAıNTAıNERS: CHANGES ON THE SALIVARY pH WERE MEASURED | baseline-3rd month measure assessing change
  Salivary pH was measured by pH meter (pH= -log hydrogen ion)
FOR FıXED SPACE MAıNTAıNERS: CHANGES ON THE SALIVA FLOW RATE, WERE MEASURED | baseline-3rd month measure assessing change
  Saliva flow rate was computed in ml/ min
FOR FıXED SPACE MAıNTAıNERS: CHANGES ON THE SALIVARY STREPTOCOCCUS MUTANS COUNTS WERE MEASURED | baseline-3rd month measure assessing change
  Strep. mutans were counted by numbers of colony-forming units (CFU) per ml (milliliter)
FOR FıXED SPACE MAıNTAıNERS: CHANGES ON THE SALIVARY LACTOBACILLUS COUNTS WERE MEASURED | baseline-3rd month measure assessing change
  Lactobacilli were counted by numbers of colony-forming units (CFU) per ml (milliliter)
FOR FıXED SPACE MAıNTAıNERS: CHANGES ON THE SALIVARY pH WERE MEASURED | baseline-6 th month measure assessing change
  Salivary pH was measured by pH meter (pH= -log hydrogen ion)
FOR FıXED SPACE MAıNTAıNERS: CHANGES ON THE SALIVARY FLOW RATE WERE MEASURED | baseline-6 th month measure assessing change
  Saliva flow rate was computed in ml/ min
FOR FıXED SPACE MAıNTAıNERS: CHANGES ON THE SALIVARY STREPTOCOCCUS MUTANS COUNTS WERE MEASURED | baseline-6 th month measure assessing change
  Strep. mutans were counted by numbers of colony-forming units (CFU) per ml (milliliter)
FOR FıXED SPACE MAıNTAıNERS: CHANGES ON THE SALIVARY LACTOBACILLUS COUNTS WERE MEASURED | baseline-6 th month measure assessing change
  Lactobacilli were counted by numbers of colony-forming units (CFU) per ml (milliliter)
FOR REMOVABLE SPACE MAıNTAıNERS: CHANGES ON THE SALIVARY pH WERE MEASURED | baseline-1st month measure assessing change
  Salivary pH was measured by pH meter (pH= -log hydrogen ion)
FOR REMOVABLE SPACE MAıNTAıNERS: CHANGES ON THE SALIVARY FLOW RATE WERE MEASURED | baseline-1st month measure assessing change
  Saliva flow rate was computed in ml/ min
FOR REMOVABLE SPACE MAıNTAıNERS: CHANGES ON THE SALIVARY STREPTOCOCCUS MUTANS COUNTS WERE MEASURED | baseline-1st month measure assessing change
  Strep. mutans were counted by numbers of colony-forming units (CFU) per ml (milliliter)
FOR REMOVABLE SPACE MAıNTAıNERS: CHANGES ON THE SALIVARY LACTOBACILLUS COUNTS WERE MEASURED | baseline-1st month measure assessing change
  Lactobacilli were counted by numbers of colony-forming units (CFU) per ml (milliliter)
FOR REMOVABLE SPACE MAıNTAıNERS: CHANGES ON THE SALIVARY pH WERE MEASURED | baseline-3rd month measure assessing change
  Salivary pH was measured by pH meter (pH= -log hydrogen ion)
FOR REMOVABLE SPACE MAıNTAıNERS: CHANGES ON THE SALIVARY FLOW RATE WERE MEASURED | baseline-3rd month measure assessing change
  Saliva flow rate was computed in ml/ min
FOR REMOVABLE SPACE MAıNTAıNERS: CHANGES ON THE SALIVARY STREPTOCOCCUS MUTANS COUNTS WERE MEASURED | baseline-3rd month measure assessing change
  Strep. mutans were counted by numbers of colony-forming units (CFU) per ml (milliliter)
FOR REMOVABLE SPACE MAıNTAıNERS: CHANGES ON THE SALIVARY LACTOBACILLUS COUNTS WERE MEASURED | baseline-3rd month measure assessing change
  Lactobacilli were counted by numbers of colony-forming units (CFU) per ml (milliliter)
FOR REMOVABLE SPACE MAıNTAıNERS: CHANGES ON THE SALIVARY pH WERE MEASURED | baseline-6 th month measure assessing change
  Salivary pH was measured by pH meter (pH= -log hydrogen ion)
FOR REMOVABLE SPACE MAıNTAıNERS: CHANGES ON THE SALIVARY FLOW RATE WERE MEASURED | baseline-6 th month measure assessing change
  Saliva flow rate was computed in ml/ min
FOR REMOVABLE SPACE MAıNTAıNERS: CHANGES ON THE SALIVARY STREPTOCOCCUS MUTANS COUNTS WERE MEASURED | baseline-6 th month measure assessing change
  Strep. mutans were counted by numbers of colony-forming units (CFU) per ml (milliliter)
FOR REMOVABLE SPACE MAıNTAıNERS: CHANGES ON THE SALIVARY LACTOBACILLUS COUNTS WERE MEASURED | baseline-6 th month measure assessing change
  Lactobacilli were counted by numbers of colony-forming units (CFU) per ml (milliliter)

IPD SHARING:
Plan to Share IPD: No